# Statistical Analysis Plan Version 2.0, 20 July 2021

## **Protocol OP-107**

**Protocol Title:** A Study of the Pharmacokinetics of Melphalan During Treatment with Melflufen and Dexamethasone in Patients with Relapsed Refractory Multiple Myeloma and Impaired Renal Function

National Clinical Trial number: NCT03639610

# **Oncopeptides AB**

## STATISTICAL ANALYSIS PLAN



PROTOCOL OP-107

A Study of the Pharmacokinetics of Melphalan During Treatment with Melflufen and Dexamethasone in Patients with Relapsed Refractory Multiple Myeloma and Impaired Renal Function

**Protocol code:** OP-107

**SAP Version:** FINAL v2.0 **SAP Date:** 20JUL2021

**Author:** Senior Statistician, PSI CRO

Review Status: FINAL Version: 2.0 Version Date: 20JUL2021

# **DOCUMENT HISTORY**

## **VERSION HISTORY**

| Version # | Version Date |
|-----------|--------------|
| V1.0 | 21APR2021 |
| V2.0 | 20JUL2021 |

## **REVISION HISTORY**

| Version # | Chapter | Revision Summary | Reason(s) for Revision |
|---|---|---|---|
| V1.0 | N/A | Initial release | N/A |
| V2.0 | 7.9.3<br>Laboratory<br>Data | Added "Lipegfilgrastim" in the list of coded preferred term for defining G-CSF for analysis. | The coded preferred term,<br>"Lipegfilgrastim" should be<br>considered G-CSF for analysis. |
| | | Added eGFR for analysis using toxicity grades. | This is to summarize eGFR toxicity grade data available. |
| | 7.9.2 Adverse<br>Events | Remove the clause regarding death before the start of subsequent anticancer treatment for the summary of death. | This is to summarize all death in a table regardless of the timing of the subsequent anticancer treatment started. |
| | 7.9.7 Chest x-ray | Added a section of chest x-ray. | This is to document chest x-ray data by a listing. |


## **APPROVAL SIGNATURES**

**STUDY TITLE:** A Study of the Pharmacokinetics of Melphalan During Treatment with Melflufen and Dexamethasone in Patients with Relapsed Refractory Multiple Myeloma and Impaired Renal Function

**PROTOCOL NUMBER:** OP-107 v.5.0. (Amendment 4 dated January 22, 2021)

**SAP** FINAL v2.0, July 20, 2021 PSI Author: Senior Statistician Signature: Date: ..... ..... Peer-reviewer Statistician: Senior Group Leader Biostatistics Signature: Date: ..... ..... Project Manager: Signature: Date: ..... ..... Medical Writer: Signature: Date: ..... ..... Oncopeptides AB Study Statistician: Signature: Date: ..... ..... Clinical Study Physician: Signature: Date: ..... Head of Clinical Pharmacology and Translational Science: Signature: Date: ..... .....


# **TABLE OF CONTENTS**

## Contents

| LIST | OF AE | BREVIATIONS | 6 |
|---|---|---|---|
| 1. | INTR | ODUCTION | 8 |
| 2. | STUE | OY OBJECTIVE | 8 |
| | 2.1 | Primary Objectives | 8 |
| | 2.2 | Secondary Objectives | 8 |
| | 2.3 | Exploratory Objectives | 9 |
| 3. | STUE | DY DESCRIPTION | 9 |
| | 3.1 | Study Design | 9 |
| | 3.2 | Study Treatment | |
| | 3.3 | Data and Safety Monitoring Committee | 0 |
| 4. | SAME | PLE SIZE AND POWER CALCULATION1 | 1 |
| 5. | ANAL | YSIS ENDPOINTS1 | 1 |
| | 5.1 | Primary Endpoints | 1 |
| | 5.2 | Secondary Endpoints | .1 |
| | 5.3 | Exploratory Endpoints | .1 |
| 6. | ANAL | YSIS POPULATIONS1 | 2 |
| 7. | ANAL | YTICAL PLAN AND STATISTICAL METHODS1 | 2 |
| | 7.1 | General Conventions and Statistical Considerations | 2 |
| | 7.2 | Definition of Baseline, Study Visits, and Visit Windows | .3 |
| | 7.3 | Handling of Missing Data1 | 4 |
| | 7.4 | Patient Disposition | 6 |
| | 7.5 | Protocol Deviations | |
| | 7.6 | Patient Characteristics | |
| | | 7.6.1 Baseline and Demographic Characteristics | |
| | | 7.6.3 Multiple Myeloma Disease History | |
| | | 7.6.4 Prior MM Therapies | |
| | <b>-</b> - | 7.6.5 Prior and Concomitant Medication | |
| | 7.7 | Pharmacokinetics Analysis | |
| | 7.8 | Efficacy Endpoints and Analysis | |
| | | 7.8.2 Time to Event Parameters | 8 |
| | | 7.8.3 Efficacy Assessments | |
| | 7.9 | Safety Endpoints and Analysis | |
| | | 7.9.1 Exposure to Study Treatment | |
| | | 7.9.3 Laboratory Data3 | 35 |
| | | 7.9.4 Vital Signs | |
| | | 7.9.5 Physical Examination | Ø |

Review Status: FINAL Version: 2.0

Version Date: 20JUL2021

| | | 7.9.6 | 12-lead Electrocardiogram (ECG) | 38 |
|-----|------|---------|--------------------------------------------|----|
| | | 7.9.7 | Chest X-Ray | 38 |
| | 7.10 | | Indpoints and Analysis | |
| | | 7.10.1 | ĖCOG | 38 |
| | | 7.10.2 | eGFR | 38 |
| 8. | INTE | RIM ANA | ALYSIS | 39 |
| 9. | DEV | ATIONS | FROM ANALYSIS AS DESCRIBED IN THE PROTOCOL | 39 |
| 10. | PRO | GRAMMI | ING SPECIFICATION | 39 |
| 11. | REF | ERENCE | s | 39 |


## **LIST OF ABBREVIATIONS**

| | BREVIATIONS |
|---|---|
| AE | adverse event |
| ALT | alanine aminotransferase |
| ANC | absolute neutrophil count |
| AST | aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| AUC | area under curve |
| $AUC_{(0-\infty)}$ | area under the concentration-time profile from 0 hours to infinity |
| $AUC_{(0-t)}$ | area under the concentration-time profile from 0 hours to the last |
| | measurable concentration |
| CB | clinical benefit |
| CBR | clinical benefit rate |
| CKD-EPI | chronic kidney disease epidemiology collaboration |
| CI | confidence interval |
| cm | centimeters |
| CR | complete response |
| CTCAE | common terminology criteria for adverse events |
| CV% | coefficient of variation |
| DOCB | duration of clinical benefit |
| DOR | duration of response |
| DSMC | Data Safety Monitoring Committee |
| ECG | electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | electronic case report form |
| eGFR | estimated glomerular filtration rate |
| EMD | extramedullary disease |
| EOT | end of treatment |
| FISH | fluorescence in situ hybridization |
| FLC | free light chain |
| ICH | International Council for Harmonisation |
| IFE | immunofixation |
| Ig | immunoglobulin |
| IMiD | immunomodulatory drug |
| IMWG | International Myeloma Working Group |
| IMWG-URC | International Myeloma Working Group Uniform Response Criteria |
| ISS | International Staging System |
| K-M | Kaplan-Meier |
| LDH | lactate dehydrogenase |
| LLOQ | lower limit of quantification |
| mAb | monoclonal antibodies |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | milligrams |
| ml | milliliter |
| MM | multiple myeloma |
| 1/11/1 | moniple injereniu |


| MR | minimal response |
|------------------|-----------------------------------------------------------|
| NCA | non-compartmental analysis |
| NCI | National Cancer Institute |
| NDA | New drug application |
| ORR | overall response rate |
| OS | overall survival |
| PD | progressive disease |
| PFS | progression free survival |
| F-U | follow-up |
| PI | proteasome inhibitor |
| PK | pharmacokinetic(s) |
| PR | partial response |
| PT | preferred Term |
| R-ISS | revised international staging system |
| RRMM | relapsed refractory multiple myeloma |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| sCR | stringent complete response |
| S-Cr | serum creatinine |
| SD | standard deviation; stable disease (depending on context) |
| SDG | standardized drug groupings |
| SDTM | study data tabulation model |
| SFLC | serum free light chain |
| SMQ | standardized MedDRA query |
| SOC | system organ class |
| SPEP | serum protein electrophoresis |
| t <sub>1/2</sub> | elimination half-life |
| TEAE | treatment-emergent adverse event |
| TTR | time to response |
| ULN | upper limit of the normal range |
| UPEP | urine protein electrophoresis |
| VGPR | very good partial response |
| WBC | white blood cells |
| WHO | World Health Organization |
| WHODD | World Health Organization Drug Dictionary |

## 1. INTRODUCTION

This statistical analysis plan (SAP) describes the statistical analysis and reporting for the study protocol OP-107 v.5.0. (Amendment 4 dated January 22, 2021) entitled; A Study of the Pharmacokinetics of Melphalan During Treatment with Melflufen and Dexamethasone in Patients with Relapsed Refractory Multiple Myeloma and Impaired Renal Function. The purpose of the plan is to outline the types of analyses and data presentations that will address the study objectives outlined in the protocol, and to explain in detail how the data will be handled and analyzed, adhering to commonly accepted standards and practices of biostatistical analysis in the pharmaceutical industry. If the protocol is amended, this SAP will be revised as required. The plan will be finalized before the study database is locked.

The statistical principles applied in the design and planned analyses of this study are consistent with International Council for Harmonisation (ICH) guidelines E9 (Statistical Principles for Clinical Trials).

This SAP does not include the description of the population pharmacokinetic (PK) modeling analysis, which is described in a separate analysis plan.

## 2. STUDY OBJECTIVE

## 2.1 PRIMARY OBJECTIVES

- To evaluate the relationship between renal function and the PK parameters for melphalan during treatment with melflufen
- To assess the safety and tolerability of melflufen in patients with moderate (Cohort 1a and 1b) and severe (Cohort 2a and 2b) renal impairment

## 2.2 SECONDARY OBJECTIVES

- To assess the best tumor response as well as overall response rate (ORR)
- To assess the progression free survival (PFS)
- To assess duration of response (DOR) in patients with ≥ partial response (PR) (stringent complete response (sCR), complete response (CR), very good partial response (VGPR), PR) as best response


• To assess clinical benefit rate (CBR) and duration of clinical benefit (DOCB) (i.e., proportion of patients with ≥ minimal response (MR)) as best response

• To assess time to response (TTR) in patients with a PR or better and time to clinical benefit (CB) for patients with MR or better

• Overall Survival (OS)

### 2.3 EXPLORATORY OBJECTIVES

• To assess changes in renal function

### 3. STUDY DESCRIPTION

## 3.1 STUDY DESIGN

This multicenter study will enroll patients with relapsed refractory multiple myeloma (RRMM) following 2-4 lines of prior therapy.

Patients will be treated with melflufen 10-40 mg on Day 1 and dexamethasone 40 mg on Days 1, 8, 15 and 22 of each 28-day cycle. Patients  $\geq$  75 years of age will have a reduced dose of dexamethasone of 20 mg on Days 1, 8, 15 and 22.

### 3.2 STUDY TREATMENT

There are four Cohorts in the study: 1a, 1b, 2a and 2b.

Cohort 1a (estimated glomerular filtration rate [eGFR] of ≥ 30 ml/min to < 45 ml/min):
 <p>Patients will be treated with Melflufen 40 mg on Day 1 and dexamethasone 40 mg on Days
 1, 8, 15 and 22 of each 28-day cycle.

Following approval of Amendment 2, Cohort 1a will close for enrollment and Cohort 1b will open for a minimum of 6 additional patients.

• Cohort 1b (eGFR of ≥ 30 ml/min to < 45 ml/min): Patients will be treated with Melflufen 30 mg on Day 1 and dexamethasone 40 mg on Days 1, 8, 15 and 22 of each 28-day cycle.

Cohort 2a will only open if recommended by Data Safety Monitoring Committee (DSMC) after evaluating data from Cohort 1a and 1b.


• Cohort 2a (eGFR of  $\geq$  15 ml/min to  $\leq$  30 ml/min): Patients will be treated with melflufen

20 mg (recommended dose by DSMC) on Day 1 and dexamethasone 40 mg on Days 1, 8,

15 and 22 of each 28-day cycle.

Cohort 2b will only open if recommended by DSMC after evaluating data from Cohort 1a, 1b and

2a.

• Cohort 2b (eGFR of  $\geq$  15 ml/min to  $\leq$  30 ml/min): Patients will be treated with melflufen

30 mg on Day 1 and dexamethasone 40 mg on Days 1, 8, 15 and 22 of each 28-day cycle.

Patients ≥ 75 years of age will have a reduced dose of dexamethasone of 20 mg on Days 1, 8, 15

and 22. Patients will be assessed for response after each cycle according to the International

Myeloma Working Group Uniform Response Criteria (IMWG-URC) (Rajkumar, 2011). Patients

may continue treatment until there is documented disease progression, unacceptable toxicity or the

patient/treating physician determines it is not in the patient's best interest to continue.

Dose modifications and delays in therapy may be implemented based on patient tolerability as

detailed in the protocol. In the event of a cycle delay, unrelated to dexamethasone toxicity, it is

recommended to continue dexamethasone weekly.

3.3 DATA AND SAFETY MONITORING COMMITTEE

An independent DSMC will perform surveillance of efficacy/safety balance at regular intervals

and on as needed basis during the study and assess the benefit/risk profile of the study, to safeguard

the interest of study participants. The DSMC will consist of lead CRO global medical monitor

investigator and Sponsor representative(s) and headed by an independent chairperson.

All reported grade 3-4 treatment-related non-hematological adverse events (AEs), as well as all

serious adverse events (SAEs), and any treatment-related deaths due to hematologic or non-

hematologic AEs, as well as efficacy and PK data will then be presented to the DSMC.

Cohort 2 will only be initiated following DSMC review of the PK and safety profile of at least 6

patients in Cohort 1. If the DSMC advises to proceed with Cohort 2, at least 6 patients with eGFR

≥ 15 ml/min to < 30 ml/min will be enrolled and analyzed for safety and PK data. The DSMC will

advise if Cohort 2 should continue as planned. Cohort 2 will have two parts, Cohort 2a and 2b.

After at least 6 patients in Cohort 2a with eGFR ≥ 15 ml/min to < 30 ml/min have been evaluated,

CONFIDENTAL 


the DSMC may advise if a higher starting dose (Cohort 2b, 30 mg melflufen) should be investigated.

If the DSMC considers the benefit/risk profile different from previous knowledge of efficacy and safety the DSMC may recommend change to the protocol, additional safety monitoring or stopping further recruitment.

All activities and processes surrounding the DSMC will be outlined in the DSMC charter.

## 4. SAMPLE SIZE AND POWER CALCULATION

Enrollment of approximately 35 PK evaluable patients is considered sufficient for a reliable assessment of the PK parameters, at least 6 patients per cohort.

## 5. ANALYSIS ENDPOINTS

### 5.1 PRIMARY ENDPOINTS

- PK parameters of melphalan
- Frequency and grade of AE's

## 5.2 SECONDARY ENDPOINTS

- ORR
- CBR
- PFS
- DOR
- DOCB
- TTR
- Best response during the study (sCR, CR, VGPR, PR, MR, stable disease (SD) or progressive disease (PD))
- OS

## 5.3 EXPLORATORY ENDPOINTS

7 Review Status: FINAL Version: 2.0


• Renal function: The level of eGFR determined at baseline and the start of each cycle

6. ANALYSIS POPULATIONS

Safety Analysis Set

The safety analysis set is defined as all patients who received at least one or partial dose of

melflufen or dexamethasone. The safety analysis set will be the primary population for the

summaries of all exposure, efficacy and safety data. Demographics and disposition data will also

be summarized based on the safety analysis set.

All listings will be presented based on the safety analysis set.

**PK Analysis Set** 

All patients that have received at least one melflufen dose and have sufficient PK samples taken

after this infusion (three samples as scheduled post-infusion), i.e. patients with at least one

treatment cycle with three measurable melphalan concentrations within the same cycle.

This analysis set will be used for the PK analysis.

**Efficacy Analysis Set** 

All patients that complete 2 doses of melflufen and have relevant baseline and follow-up disease

assessments after the second dose of melflufen. This analysis set will be used for sensitivity

analysis of all the efficacy parameters.

Relevant disease assessments: Serum protein electrophoresis (SPEP), urine protein electrophoresis

(UPEP), serum free light chain (SFLC), and immunofixation (IFE) in serum and urine.

Note: All of these relevant lab parameters at different timepoints will be considered for follow-up

disease assessments as long as taken after the second dose of melflufen.

7. ANALYTICAL PLAN AND STATISTICAL METHODS

7.1 GENERAL CONVENTIONS AND STATISTICAL CONSIDERATIONS

All statistical analyses will be performed using SAS statistical analysis software (SAS,

SAS/GRAPH and SAS/STAT; version 9.4 or higher of SAS for Windows [SAS Institute Inc.;

Cary, NC, USA]).

CONFIDENTAL 

Review Status: FINAL

Version: 2.0


Descriptive statistics for continuous variables will include the number of patients with non-missing

data (n), arithmetic mean, standard deviation (SD), median, minimum and maximum. Summary

statistics for categorical variables will contain count and percentage based on the number of

patients in the selected analysis population. Percentages will be presented to one decimal, except

for zero and one hundred percent, which will be presented as 0% and 100% respectively.

For descriptive statistics of continuous variables, the accuracy of the minimum and maximum and

should match the original data, for the mean and median one more decimal point in addition to the

original data will be presented, and for SD two more decimal points in addition to the original data

will be presented. For the derived variables (e.g., time since diagnosis) minimum and maximum

will be presented with one decimal after point; mean, median and SD will be applied following

the rule above. Presented decimal places should however not be greater than 4.

For PK descriptive statistics significant figures will be used for precision: mean, geometric mean

and median values are shown with 4 significant figures, and standard deviation and CV% with 3

significant figures.

Any data categorization will be done based on the original data, before rounding is applied.

Unless otherwise specified, the denominators for the percentages will be based on the number of

patients with non-missing data in the population used in each column. For the summaries presented

by time points, the denominator will be the number of patients with non-missing data at each time

point. A "missing" category will be included for any parameter for which information is missing,

without a percentage.

By default the data collected in the electronic case report form (eCRF) and by external vendors

will be used for analysis unless it is specified that additional derivation is required.

There will be no formal statistical analysis in this study. Results will be presented using descriptive

statistics by cohort (Cohort 1a, Cohort 1b, Cohort 2a and Cohort 2b) and overall.

For treated patients all data collected will be presented in the listings. Some derived parameters

will also be presented in the listings: i.e. derived international staging system (ISS) and revised

international staging system (R-ISS), cytogenetics abnormalities risk-level, best confirmed

response during the study, and PK parameters.

7.2 DEFINITION OF BASELINE, STUDY VISITS, AND VISIT WINDOWS

Review Status: FINAL

Version: 2.0


In general the baseline is the last available assessment prior to the first dose of study drug (the

earliest of melflufen and dexamethasone start date).

Where assessments are made on the day of first treatment and the time is available for comparison,

the time should be used to recognize whether or not the assessment was prior to the first treatment

and thus should be used as a baseline. If only the date is in place and time is not available, for

assessments on the day of first treatment that are per protocol scheduled to take place prior to

treatment, it will be assumed that the assessment is pre-dose, and is a valid baseline assessment.

Refer to the protocol for the study visit schedule.

Note that for this study there is no study day 0, so the day immediately prior to study day 1 is study

day -1. For any events on or after the first dose of study drug, study day is calculated as: event date

– date of first administration of study treatment + 1. As such, the first dose date was study day 1.

For any events before the first dose date, study day is calculated as: event date - date of first

administration of study treatment. As such, one day before first dose date was study day -1.

Because unscheduled assessments are not associated with any scheduled time point, they are

excluded from all summaries by time point. Unscheduled visits will be considered for the baseline

values derivations. Unscheduled assessments will be considered when deriving myeloma response

parameters as described in the Section 7.7 and for analysis of laboratory parameters by worst

toxicity grade as specified in the Section 7.8.3 of this SAP. All unscheduled assessments will be

presented in the respective listings.

The data will be analyzed according to the visits recorded in the eCRF and no analysis windows

will be applied.

7.3 HANDLING OF MISSING DATA

If only a partial date is available and is required for a calculation (e.g., time since diagnosis, time

since most recent relapse, determination of whether a medication is concomitant or an AE is

treatment-emergent), the following standards will be applied:

• Start dates (e.g., AE onset date or start date of medication, date of diagnosis, date of

relapse). For missing start day only - day will be imputed as the first day of the month (i.e.,

1) with the following exception: if the partial date falls in the same month and year as the

date being used in the calculation (e.g., first dose date, informed consent date), then the

CONFIDENTAL

Review Status: FINAL

Version: 2.0


partial date will be imputed to equal the date being used for the calculation, unless there is

a complete end date which is earlier.

For missing start day and month - day and month will be imputed as the first day of the

year (i.e., 01 January) with the following exception: if the partial date falls in the same year

as the date being used in the calculation (e.g., first dose date, informed consent date), then

the partial date will be imputed to equal the date being used for the calculation, unless there

is a complete end date which is earlier.

• Stop dates (e.g., AE resolution date or stop date of medication). For missing stop day only

- day will be imputed as the last day of the month (i.e., 28, 29, 30, or 31).

• For missing stop day and month - day and month will be imputed as the last day of the year

(i.e., 31 December).

Any partial dates will be displayed in data listings without imputation of missing days and/or

months (e.g., MAR2011, 2009).

In case of incomplete date of relapse, for the purpose of calculation of the time since most recent

relapse, the rules mentioned above for the partial start date will be used. However, for the date of

frontline transplant in calculation of time since frontline transplant to relapse and for the date of

relapse in derivation of refractory status, the simplified approach of assigning first day of a month

in case of missing day and 01 January in case of missing month and day will be used. This simple

approach will be also applied to impute the partial date of relapse in the calculation of time since

the frontline transplant to relapse with the following exception in order to avoid yielding a negative

duration due to imputation: The partial date of relapse will be imputed to the date of frontline

transplant in case the partial date falls in the same month and year (if only day is missing) or in the

same year (if day and month are missing).

If time is not available but is required for a calculation (e.g., timing of AE vs study drug

administration), the most conservative approach should be used, i.e. assuming that the time of AE

was after study drug administration or that the time of concomitant medication was after AE.

AEs with missing relationship are considered related for the purposes of summaries. In case of

multiple cases, the information regarding the number of imputed relationships will be provided in

the footnote of the respective summaries.

AEs with missing severity are considered severe (grade 3) for the purposes of summaries. Imputed


relationship and severity will not be included in the listings.

eGFR will be derived using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula (See Section 7.6.3) if eGFR is not reported but serum creatinine is available for the corresponding visit.

The handling of dropouts and missing disease status assessments for the efficacy variables is described in their definitions in the relevant sections.

### 7.4 PATIENT DISPOSITION

Disposition summary will be based on the safety analysis set and presented by cohort and overall. The disposition of patients includes:

- Number (%) of patients in safety, PK and efficacy analysis sets
- Number (%) of patients permanently discontinued from the treatment along with the primary reasons for permanent treatment discontinuation
- Number (%) of death reported up to the end of treatment visit
- Number (%) of patients who had PFS follow-up (F-U) and by the following categories using counts and percentages based on the number of patients who had PFS F-U
  - o Progressive disease (PD) and confirmed PD
  - o Diagnosed with a second primary malignancy
  - Started subsequent therapy
- Number (%) of patients who had OS F-U and by the following categories using counts and percentages based on the number of patients who had OS F-U
  - o Diagnosed with a second primary malignancy
  - Started subsequent therapy
  - o Survival status at the last OS-FU
- Number (%) of patients discontinued from the study and reasons for study discontinuation Treatment discontinuations due to AE specific to COVID-19 or other pandemic-related reasons will be presented separately.

All patient disposition information will be presented in the respective listings.

### 7.5 Protocol Deviations

Major protocol deviations will be summarized by the deviation type for the safety analysis set by cohort and overall. All protocol deviations will also be provided in a listing. Separate listings for major protocol deviations, COVID-19 pandemic-related protocol deviations, and major COVID-19 pandemic-related protocol deviations will also be provided.

#### 7.6 PATIENT CHARACTERISTICS

#### 7.6.1 BASELINE AND DEMOGRAPHIC CHARACTERISTICS

The following demographic and baseline characteristics will be summarized descriptively for the safety analysis set by cohort and overall:

- Age (years)
- Age categories (<65,  $\ge 65$  to  $\le 75$ , >75)
- Sex
- Race
- Ethnicity
- Baseline fertility status
- Baseline height (cm)
- Baseline weight (kg)
- Baseline Eastern Cooperative Oncology Group (ECOG) performance status

A listing will be provided for patient's demographic and baseline characteristics.

Separate listings will be provided for pregnancy test and ECOG results.

#### 7.6.2 MEDICAL HISTORY AND CURRENT MEDICAL CONDITIONS

Medical history will be summarized by Medical Dictionary of Regulatory Activities (MedDRA) (version 24.0 or higher), System Organ Class (SOC) and preferred term (PT) using number (n) and percentage (%) of patients having at least one occurrence of a disease for the safety analysis set by cohort and overall. Any medical history of COVID-19 will be presented as separate PTs specific to COVID-19 or SARS-CoV-2.

A listing will be provided for patient medical history.

#### 7.6.3 MULTIPLE MYELOMA DISEASE HISTORY

The following disease characteristics at diagnosis will be summarized descriptively for the safety analysis set by cohort and overall:


- Stage of disease (ISS and R-ISS)
- Heavy chain and light chain subtypes
- Evidence of lytic bone disease
- Evidence of extramedullary disease (EMD)

The following disease characteristics at baseline/study entry will be summarized descriptively for the safety analysis set by cohort and overall:

- Stage of disease (ISS and R-ISS), eCRF reported and derived (see Table 1.)
- Heavy chain and light chain subtypes
- Evidence of lytic bone disease
- Evidence of EMD
- Disease status
- Time since diagnosis in years (calculated as [date of first dose of study drugs (the earliest of melflufen and dexamethasone first dose) date of diagnosis+1]/365.25). Partial dates will be imputed according to the section 7.3 of this SAP
- Time since most recent relapse/progression in months (calculated as [date of first dose of study drugs (the earliest of melflufen and dexamethasone first dose) date of most recent relapse/progression+1]/30.4375)
- Baseline SPEP, UPEP, kappa/lambda values; For descriptive statistics, in case of the second SPEP value being available as >0 g/L, the SPEP value will be derived as follows; Otherwise, in case of the second SPEP value being 0 g/L or not available, descriptive statistics will be produced without considering the second SPEP.
  - o If there are more than one heavy chain subtypes (IgG, IgA, IgD, IgE, IgM) at study entry, the worst/higher values between the two available SPEP values will be used for descriptive statistics.
  - o If there is only one heavy chain subtype (IgG, IgA, IgD, IgE, IgM) at study entry, the sum of the two available SPEP values will be used for descriptive statistics.
- Baseline maximum bone marrow plasma cells involvement (%) as values and by categories (<30%, ≥30 to <60%, ≥60%) (Note: The maximum bone marrow plasma cells involvement will be defined as the highest value amongst any of the available test results from the following bone marrow lab parameters: plasma cells ratio from bone marrow test, immature plasma cells/total cells based on bone marrow biopsy test or bone marrow aspiration/differential test.)
- Laboratory assessments
  - O Baseline β2 microglobulin (mg/L) as continuous values and categories ( $< 3.5, \ge 3.5$  to < 5.5 and > 5.5)

- O Baseline platelet count  $(10^9/L)$  as continuous values and categories  $(<75, \ge 75 \text{ to} \le 100, >100 \text{ to} \le 150, >150)$
- O Baseline absolute neutrophil count (ANC) ( $10^9/L$ ) as continuous values and categories ( $<1.0, \ge 1.0$  to  $\le 1.5$ , and >1.5)
- Baseline hemoglobin (g/L) as continuous values and categories ( $<80, \ge80$  to  $\le100, >100$ )
- o Baseline lactate dehydrogenase (LDH) (u/L) as continuous values and categories (<1.5xULN and ≥1.5xULN)
- Baseline albumin (g/L) as continuous values and categories ( $<35, \ge35$ )
- Baseline creatinine as continuous values
- O Baseline eGFR (mL/min/1.73m2) as continuous values and categories ( $< 15, \ge 15$  to  $< 30, \ge 30$  to  $< 45, \ge 45$ )
- Screening eGFR (mL/min/1.73m2) as continuous values and categories (< 15, ≥15 to <30, ≥30 to <45, ≥45) (Note: The latest available screening value (including unscheduled if available) will be used for analysis.)</li>
- Baseline corrected calcium as continuous values

For patients for whom only creatinine clearance was calculated at baseline as a basis for enrolment values for renal function will be recalculated as eGFR using CKD-EPI formula:

$$eGFR = 141 * min(Scr/\kappa, 1)^{\alpha} * max(Scr/\kappa, 1)^{-1.209} * 0.993^{Age} * 1.018 [if female] * 1.159 [if black]$$

\*Scr is serum creatinine (mg/dL),  $\kappa$  is 0.7 for females and 0.9 for males,  $\alpha$  is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/ $\kappa$  or 1, and max indicates the maximum of Scr/ $\kappa$  or 1.

In addition to the above, ISS Stage and Revised ISS (R-ISS) Stage will be derived at study entry [Palumbo, 2015], (see Table 1).

ISS will be derived from screening serum  $\beta 2$  microglobulin and screening albumin. This derived ISS will in turn be used with screening serum LDH and high-risk cytogenetics at study entry as defined by the R-ISS guidelines to derive R-ISS. Derived ISS and R-ISS will be referred as "Derived ISS" and "Derived R-ISS" respectively. (Note: This derivation will consider the latest available screening value for  $\beta 2$  microglobulin, albumin, and serum LDH (including unscheduled if available).


Table 1: Standard Risk Factors for MM and the Revised ISS (R-ISS)

| Standard Risk Factors for MM and the Revised ISS (R-ISS) | |
|---|---|
| Prognostic Factor | Criteria |
| ISS Stage | |
| Stage I | Serum B2-microglobulin < 3.5 mg/L, serum albumin ≥ 3.5 g/dL |
| Stage II | Not ISS stage I or III |
| Stage III | Serum B2-microglobulin ≥ 5.5 mg/L |
| Chromosomal abno | rmalities (CA) by interphase florescent in situ hybridization (iFISH) |
| High-Risk | Presence of del(17p) and/or translocation of t(4:14) and/or translocation of t(14:16) |
| Standard-Risk | ındard-Risk No high-risk CA |
| Lactate Dehydroger | nase (LDH) |
| Normal Serum LDH =< upper limit of normal (ULN) | |
| High | Serum LDH > ULN |
| A new model for risk stratification of MM R-ISS | |
| Stage I | ISS stage I and standard-risk CA by iFISH and normal LDH |
| Stage II | Not R-ISS stage I or III |
| Stage III ISS stage III and either high-risk CA by iFISH or LDH | |

A separate summary dedicated to cytogenetics investigations at diagnosis and study entry will be presented, including type of cytogenetic analysis (iFISH, karyotype), and the number and percentage of patients having particular types of cytogenetic abnormalities. Cytogenetics abnormalities at study entry will also be pooled by risk level (high-risk, standard-risk and unknown) as follows depending on the type of cytogenetic analysis:

- High-risk based on iFISH is defined in case the following abnormalities were found: deletion (17p), gain 1q (+1q), gain (1q21); t (4;14), t(4;14) (p16;q32), t (14;16), t (14;16) (q32;q23), t(14;20), t(14;20) (q32;q11).
- Standard-risk based on iFISH consists of patients who have a genetic subtype recorded but none of the genetic subtypes categorized as high-risk based on iFISH.
- Unknown: consists of patients for whom the iFISH procedure was not done or unevaluable.
- High-risk based on karyotype is defined in case the following abnormalities were found: deletion (13) or deletion (13q).
- Standard-risk based on karyotype consists of patients who have a genetic subtype recorded but none of the genetic subtypes categorized as high-risk based on karyotype.


• Unknown: consists of patients for whom the karyotype procedure was not done or

unevaluable.

Bone lesion assessments at screening will be analyzed descriptively with the number and percent

of patients, including the number and percent of patients for whom skeletal survey was performed,

method of skeletal survey, result of exam, bone lesions locations. The same information will be

presented for the other imaging procedures.

Listings will be provided for MM history, bone lesion assessments and bone marrow aspirate.

7.6.4 PRIOR MM THERAPIES

The following information related to prior MM therapies will be summarized for the safety

analysis set by cohort and overall:

• Number and percentage of patients who had a transplant.

• Number of patients who had a salvage transplant (defined as any transplant where the

patient has already had one or more transplants in earlier lines). Planned tandem autologous

or autologous-allogeneic are considered as one transplant.

• Frontline transplant type (allogeneic or autologous); Frontline transplant is the first

transplant per patient irrespective in which therapy line it was applied. The number and

percentage of patients having frontline transplant per prior therapy line will be presented.

• Number and percentage of patients with the tandem transplant.

• Number and percentage of patients with at least one prior autologous transplant, and

number and percentage of patients with two or more prior autologous transplants

• Number of prior autologous transplants

• Time from frontline transplant to the earliest relapse following frontline transplant (not

necessarily after the prior therapy line when frontline transplant occurred) in years (as

continuous variable as well as per categories < 1 year,  $\ge 1$  year to < 1.5 years,  $\ge 1.5$  years to

≤2 years, >2 years; To be calculated as [date of earliest relapse following the frontline

transplant – date of frontline transplant +1]/365.25. Partial dates will be imputed according

to the section 7.3 of this SAP)

• Number of prior systemic therapy lines

• Best response to the last prior line of systemic therapy

CONFIDENTAL 


• Refractory status to the last prior line of systemic therapy

• Number and percentage of patients with any prior lines including: immunomodulatory

drugs (IMiD's), proteasome inhibitors (PI's), alkylators, anti-CD38 monoclonal antibodies

(mAb), other mAb and others

• Number and percentage of patients receiving any of above agents in the last prior line.

• The number and percentage of patients refractory to any of the above agents in at least one

prior regimen

• The number and percentages patients refractory to any of the above agents in the last prior

line

• Number and percentage of patients who received IMiD and PI (double-class) in any of

prior lines of therapies

• Number and percentage of patients, double refractory to PI and IMiD in any of prior lines

of therapies);

• Number and percentage of patients who received IMiD, PI, and anti-CD38 mAb (triple-

class) in any of prior lines of therapies

• Number and percentage of patients, that are refractory and/or intolerant to a PI, an IMiD,

and an Anti-CD38 mAb (Triple class refractory) in any of prior lines of therapies.

Intolerance is defined when a patient stopped treatment due to toxicity, and as well as did

not receive a drug in the same therapeutic drug class again prior to entering the current

study.

Number and percentage of patients with prior radiotherapy

The next list of drugs is associated with each drug class using World Health Organization Drug

Dictionary (WHODD) version March 2021 or higher:

• IMiD is defined as WHODD Standardized Drug Groupings (SDG) "Antineoplastic

thalidomide analogues"

• PI is defined as WHODD SDG "Antineoplastic proteasome inhibitors"

• Alkylators is defined as WHODD SDG "Antineoplastic alkylating drugs"

• Anti-CD38 mAb is defined as WHODD SDG "Antineoplastic CD38 antigen inhibitors"

• Other mAb is defined as WHODD SDG "Monoclonal antibodies – antineoplastics"

excluding SDG "Antineoplastic CD38 antigen inhibitors"

CONFIDENTAL 


• Other antineoplastic drugs for the treatment of MM will be referred to as 'Other'. Will be

identified by manual review of the drugs not included into the categories above.

Refractory is defined as non-responsive disease (achieving SD or PD as the best response) while

on therapy, or reason for termination was PD, or relapse/progression within 60 days after stop date

of treatment. A patient is to be deemed as refractory to a therapy line in case of refractory to at

least one of the agents in the therapy line whereas a patient is deemed as non-refractory to a therapy

line in case of non-refractory to all of agents in the therapy line. Otherwise, a patient's refractory

status to the therapy line will be considered unknown.

All patient details of prior MM therapies will be presented in the respective listings.

7.6.5 PRIOR AND CONCOMITANT MEDICATION

All concomitant medications will be coded using the WHODD version March 2021 or higher.

A medication is considered prior if stopped before the date of the first dose of study drug (the

earliest of melflufen and dexamethasone start date). Concomitant medications are defined as

medications with start date or end date on or after the date of first dose of study drug and start date

within 30 days after the date of the last dose of study drug (the latest of melflufen and

dexamethasone end date) or are ongoing at the time of first dose of study drug.

The number and percentages of patients with at least one concomitant medication will be

summarized by the Anatomical Therapeutic Chemical (ATC) class (ATC 2 and ATC 4) and

preferred name. Summaries will be presented by safety analysis set by cohort and overall. Patients

may have more than one medication per ATC class and preferred name. At each level of patient

summarization, a patient is counted once if he/she reported one or more medications at that level.

The summaries will be ordered by descending frequency of ATC class and preferred name within

each ATC class in the total group. Prior medications will be presented separately in the same way.

Separate summaries will be provided for the number and percentage of patients with the following

medication categories: "Haemapoetic growth factors" (WHODD SDG "Colony stimulating

factors") and by preferred terms, as well as "Transfusions" (including next PTs: "Platelets",

"Erythrocytes").

A listing of prior and concomitant medications will be provided.

All prior and concomitant surgical/medical procedures performed within 21 days of study entry

until the EOT visit will be listed.

CONFIDENTAL 


7.7 PHARMACOKINETICS ANALYSIS

PK parameters will be calculated and provided by the Sponsor using Non-Compartmental Analysis

(NCA) and the software Phoenix WinNonlin® version 8.2 or later (Certara L.P., U.S.A.). The

following PK parameters will be assessed for melphalan.

Maximum drug concentration (C<sub>max</sub>)

C<sub>max</sub> is defined as the maximum drug concentration observed in plasma per treatment cycles

with PK sampling.

• Time of maximum concentration (T<sub>max</sub>)

Time of maximum plasma concentration  $(T_{max})$  is defined as the time at which the  $C_{max}$  occurs.

• Area under the concentration-time profile from 0 hours to the last measurable concentration

 $(AUC_{(0-t)})$ 

 $AUC_{(0-t)}$  is defined as the area under the concentration-time curve from start of dosing (time 0)

to the time of the last measured concentration. AUC<sub>(0-t)</sub> will be estimated using the Linear Up

Log Down calculation method.

• Area under the concentration-time profile from 0 hours to infinity  $(AUC_{(0-\infty)})$ 

 $AUC_{(0-\infty)}$  is defined as the total area under the concentration-time curve from start of infusion

(time 0) to the limit as the end time becomes arbitrarily large.

• Half-life (t½)

The apparent t½ is defined as the time required for the drug concentration to decrease by a

factor of one-half in the terminal phase. t½ will be estimated as ln(2) / Ke, Ke referring to

terminal phase elimination rate constant of the apparent log-linear decrease as defined by 3 data

points.

Blood samples for PK analysis of melphalan concentrations in plasma, will be collected at the

following time points:

CONFIDENTAL 


Table 4. PK sampling schedule

| | Cycle 1 and 2 |
|----------------------|--------------------------------------------------|
| Sample 1, time point | 5-10 minutes after the end of melflufen infusion |
| Sample 2, time point | 2-3 hour after the end of melflufen infusion |
| Sample 3 time point | 5-7 hours after the end of melflufen infusion |

Date and time of sample collection or reason for not being collected will be recorded in the eCRF. Concentrations and corresponding PK parameters will be provided as external files and appended to the study database.

Actual time points relative to start of melflufen infusion in minutes will be derived and used by the Pharmacokinetist for calculating parameters. Actual time in minutes will be calculated as datetime of blood sampling minus datetime of start of infusion.

All PK parameters to be calculated for melphalan are listed in Table 5. The derivation of PK parameters is done by the Pharmacokineticist. All parameters will be presented in a listing in minimum.

Table 5. PK parameters to be calculated

| Phoenix WinNonLin ID | Unit | Parameter code | CDISC submission value |
|---|---|---|---|
| Rsq | | R2 | R Squared |
| Rsq_adjusted | | R2ADJ | R Squared Adjusted |
| Corr_XY | | CORRXY | Correlation Between TimeX and Log ConcY |
| No_points_lambda_z | | LAMZNPT | Number of Points for Lambda z |
| Lambda_z | min | LAMZ | Lambda z |
| Lambda_z_int | ng/mL | LAMZINT | Lambda z Intercept |
| Lambda_z_lower | min | LAMZLL | Lambda z Lower Limit |
| Lambda_z_upper | min | LAMZUL | Lambda z Upper Limit |
| Lambda_z_span | min | LAMZSPN | Lambda z Span |
| *HL_Lambda_z | min | LAMZHL | Half-Life Lambda z |
| *Tmax | min | TMAX | Time of Cmax |
| *Cmax | ng/mL | CMAX | Max Conc |
| Cmax_D | ng/mL/mg | CMAXD | Max Conc Norm by Dose |

CONFIDENTAL 


| Tlast | min | TLST | Time of Last Nonzero Conc |
|---|---|---|---|
| Clast | ng/mL | CLST | Last Nonzero Conc |
| Clast_pred | ng/mL | CLSTP | Last Nonzero Conc Pred |
| *AUClast | min*ng/mL | AUCLST | AUC to Last Nonzero Conc |
| AUClast_D | min*ng/mL | AUCLSTD | AUC to Last Nonzero Conc Norm by Dose |
| AUCall | min*ng/mL | AUCALL | AUC All |
| *AUCINF_obs | min*ng/mL | AUCIFO | AUC Infinity Obs |
| AUCINF_D_obs | min*ng/mL/mg | AUCIFOD | AUC Infinity Obs Norm by Dose |
| AUC_%Extrap_obs | % | AUCPEO | AUC %Extrapolation Obs |
| Vss_obs | L | VSSO | Vol Dist Steady State Obs |
| Vz_obs | L | VZO | Vz Obs |
| AUCINF_pred | min*ng/mL | AUCIFP | AUC Infinity Pred |
| AUCINF_D_pred | min*ng/mL/mg | AUCIFPD | AUC Infinity Pred Norm by Dose |
| AUC_%Extrap_pred | % | AUCPEP | AUC %Extrapolation Pred |
| Vss_pred | L | VSSP | Vol Dist Steady State Pred |
| Vz_pred | L | VZP | Vz Pred |
| Cl_pred | L/min | CLP | Total CL Pred |
| AUMClast | min*min*ng/mL | AUMCLST | AUMC to Last Nonzero Conc |
| AUMCINF_obs | min*min*ng/mL | AUMCIFO | AUMC Infinity Obs |
| AUMC_%Extrap_obs | % | AUMCPEO | AUMC % Extrapolation Obs |
| AUMCINF_pred | min*min*ng/mL | AUMCIFP | AUMC Infinity Pred |
| AUMC_%Extrap_pred | % | AUMCPEP | AUMC % Extrapolation Pred |
| MRTlast | min | MRTIVLST | MRT Intravasc to Last Nonzero Conc |
| MRTINF_obs | min | MRTIVIFO | MRT Intravasc Infinity Obs |
| MRTINF_pred | min | MRTIVIFP | MRT Intravasc Infinity Pred |
| * Summarized with descriptive | etatistics as contin | mone variables and with | the geometric mean and geometric coefficient of |

<sup>\*</sup> Summarized with descriptive statistics as continuous variables and with the geometric mean and geometric coefficient of variation.

 $C_{max}$  and  $T_{max}$  will be presented with the same number of decimals as the concentration measurements and time points, while the derived PK variables will be presented with an appropriate number of significant digits based on the general practice.

It may be necessary to exclude individual PK profiles because they are erroneous or abnormal, e.g. protocol violation, documented sample handling errors etc. Such data will not be used for analysis and any excluded data should be flagged in the listings and the reason for exclusion should be documented.


Statistical methods

Descriptive statistics (arithmetic mean with corresponding SD, geometric mean with

corresponding SD, geometric coefficient of variation (CV%), median with minimum and

maximum) for drug concentrations by time point and PK variables will be provided for

melphalan.

Geometric mean and geometric CV% will be calculated as follows:

Geometric mean = GeoMean =  $exp[\{ln(y_1) + \cdots + ln(y_n)\}/n]$ ,

Geometric standard deviation =  $GeoSD = exp[SD\{ln(y_1), ..., ln(y_n)\}]$ , and

Geometric CV (%) =  $GeoCV = 100 \times \sqrt{exp\{ln(GeoSD)\}^2 - 1}$ ,

where SD is the arithmetic standard deviation.

7.8 **EFFICACY ENDPOINTS AND ANALYSIS** 

All efficacy analyses will be produced on the safety analysis set and efficacy analysis set by cohort

and overall.

All tumor response and progression-depended objectives are assessed by investigators according

to the IMWG-URC (Rajkumar, 2011).

7.8.1 RESPONSE RATES

For analysis of response rates, all percentages calculations will be based on the respective analysis

set. For analysis of the best confirmed response rates, a category of 'non-evaluable' will be added

and included in the percentage calculation for patients who cannot be categorized for the best

confirmed response (as described below). For analysis of the best unconfirmed response rates, the

same approach will be used.

**Best Overall Confirmed Response** 

Best overall confirmed response during the study, including follow-up tumor response assessments

(sCR, CR, VGPR, PR, MR, SD or PD), collected prior to the new therapy initiation, and assessed

by the investigator according to IMWG-URC, will be summarized descriptively.

Confirmed response: Two consecutive assessments with the same response result made at any

time. In case at the second consecutive assessment (made at any time) the response is higher than

**CONFIDENTAL** 


the previous one, then confirmed response (linked to the first assessment visit) will be the first one

(e.g., PR – VGPR consecutive pair will lead to a PR confirmed response at the first visit). In case

the second consecutive response is lower than the first one, then confirmed response (linked to the

first assessment visit) will be the second one (e.g. CR-VGPR consecutive pair will lead to a VGPR

confirmed response at the first visit).

**Best Unconfirmed Response** 

Defined as the best response achieved on study, i.e. a response may not be confirmed by a

consecutive assessment. Will be presented similarly to best overall confirmed response.

**Overall Response Rate** 

The ORR will be estimated as the proportion of patients who achieve a confirmed response of

sCR, CR, VGPR, or PR as their best response, as assessed by the investigator. The denominator is

the number of patients in the analysis population for particular cohort. The exact binomial two-

sided 95% confidence interval (CI) for ORR will be calculated.

**Clinical Benefit Rate** 

The CBR is the proportion of patients who achieve a confirmed minimal response or better (sCR,

CR, VGPR, PR and MR) as their best response, as assessed by the investigator. CBR will be

summarized using the same method as for ORR.

All the details of myeloma response assessment will be presented in a listing.

7.8.2 TIME TO EVENT PARAMETERS

**Progression-Free Survival** 

The PFS is defined as the time from the date of first study drug (the earliest of melflufen and

dexamethasone start date) initiation to the date of first documentation of confirmed PD or death

due to any cause, whichever occurs first. PFS time, in months, is calculated as (PFS date – date of

first study drug initiation +1)/30.4375.

Additional conventions for the PFS date derivation and censoring are defined in the Table 2 below:

CONFIDENTAL


Table 2. Conventions for PFS date derivation and censoring

| Situation | Date of Progression or Censoring | Outcome |
|---|---|---|
| No post-baseline response assessments, except in the case of death | Date of initiation of therapy (the earliest of melflufen and dexamethasone start date) | Censored |
| New anticancer therapy started<br>before documentation of PD or<br>death | Date of last response assessment prior to start of new anticancer therapy | Censored |
| Death or PD immediately after<br>more than 1 consecutively missed<br>response assessment visit* | Date of last response assessment visit without documentation of PD that is before the first missed visit | Censored |
| Unconfirmed PD as the final response assessment | Date of latest PD assessment | Progressed |
| Alive and without PD documentation | Date of last response assessment | Censored |
| Death or PD between planned response assessments | Date of death or first response assessment showing PD, whichever occurs first | Progressed |
| Death before first response assessment | Date of death | Progressed |

<sup>\*</sup>unless there was an unscheduled visit showing absence of PD between the last scheduled missing response assessment and date of PD identification

The distribution of PFS will be summarized using the Kaplan-Meier (K-M) method. The median PFS will be estimated from the 50th percentile of the corresponding K-M estimates. The 95% CI for median PFS will be constructed using the method of Brookmeyer (Brookmeyer, 1982).

K-M plots will also be produced.

A patient data listing will be provided for PFS follow-up.

## **Duration of Response (DOR)**

DOR is defined as the time in months from the first evidence of confirmed assessment of sCR, CR, VGPR, or PR to first confirmed disease progression according to the IMWG-URC or to death due to any cause. DOR is defined only for patients with a confirmed PR or better.

DOR is to be censored and summarized using the same methods as for PFS.

DOR will be derived as (DOR date – date of first documented confirmed response (≥PR) + 1)/30.4375.


**Duration of Clinical Benefit (DOCB)** 

DOCB will be calculated as time in months from the first evidence of confirmed assessment of

sCR, CR, VGPR, PR or MR to first confirmed disease progression, or to death due to any cause.

Duration of clinical benefit is defined only for patients with a confirmed MR or better. DOCB will

be censored and summarized using the same method as for PFS.

DOCB will be derived as (DOCB date – date of first documented confirmed response (≥MR) +

1)/30.4375.

Time to Response (TTR)

TTR will be calculated as time in months from first dose of study drug to first documented

confirmed response in a patient that has responded with PR or better. TTR will be presented

descriptively for patients with a response. Will be derived as (date of first documented confirmed

response ( $\geq$ PR) – date of study drug initiation +1)/30.4375.

Time to CB will be presented for confirmed response of MR or better and analyzed similarly to

TTR.

**Overall Survival (OS)** 

OS defined as time in months from date of study drug initiation to death due to any cause. Patients

still alive at the end of study, or lost to follow-up, will be censored at last day known alive. Will

be derived as (OS date – date of study drug initiation +1)/30.4375.

A patient data listing will be provided for overall survival follow-up.

7.8.3 EFFICACY ASSESSMENTS

Myeloma specific laboratory tests results, including SPEP, UPEP, serum and urine IFE, and SFLC

will be summarized descriptively by assessment visit, and this will include change from baseline

summary using descriptive statistics for continuous variables. In case the second SPEP value is

available as >0 g/L at a given time point, see the section 7.6.3 for the derivation.

All the myeloma specific laboratory tests results and other efficacy assessments (i.e.

extramedullary plasmacytoma assessment) will be presented in the listings.

CONFIDENTAL


7.9 SAFETY ENDPOINTS AND ANALYSIS

All analyses of safety will be based on the safety analysis set.

7.9.1 EXPOSURE TO STUDY TREATMENT

Exposure analysis will be based on the safety analysis set by cohort and overall.

Duration of melflufen treatment in weeks is defined as (date of last dose – date of first dose + 29

days) divided by 7.

If a patient discontinued from treatment and the end of treatment (EOT) visit happened prior to 29

days after last dose, then the duration of melflufen is defined as (date of EOT – date of first dose

+1) divided by 7.

If a patient died prior to 29 days after last dose, then the duration of melflufen is defined as (date

of death - date of first dose +1) divided by 7.

Duration of dexamethasone treatment in weeks is defined as (date of last dose – date of first

dose + 1) divided by 7.

Overall duration of treatment with study drug in weeks is defined as the longest duration of

dexamethasone or melflufen treatment.

The duration of study treatment exposure will be summarized descriptively and presented for

overall treatment duration and also separately for melflufen and dexamethasone and will include:

treatment duration in weeks, number of cycles received (and also additionally number of doses for

dexamethasone), cumulative dose (in mg) of study drug received per patient, average dose of study

drug (mg/week for melflufen and mg/week for dexamethasone), the total number and percentage

of patients receiving a dose per cycle (for overall treatment and melflufen), average duration of

infusion (min) for melflufen. Patients who received only a partial dose of melflufen for a given

cycle will be considered as having received treatment for that cycle.

Average dose of melflufen in mg/week is defined as the cumulative dose divided by the duration

of melflufen treatment (the same for dexamethasone).

Dose modification information will be summarized descriptively for any drug (melflufen and/or

dexamethasone) for overall and then also separately for melflufen and dexamethasone by cycle.

The number of patients with each action by frequency will be presented based on the

melflufen/dexamethasone administration eCRF page.

A dose delay is defined as a consecutive dose of melflufen administered on day 33 or later


following a preceding dose of melflufen (day at the moment of melflufen administration is defined

as a difference between Cycle X Day 1 (CXD1) date and C(X-1)D1 date +1). Dose delays will be

categorized as delays in weeks as 1 (day 33 to 39), 2 (day 40 to 46), 3 (day 47 to 53), 4 (day 54 to

60), and >4 weeks (day 61 or later) for each cycle.

A separate table will present the number and percentage of patients with delayed cycles for post-

cycle 1 (those with day 33 and later at the moment of melflufen administration following a

preceding dose of melflufen) as well as the number of delayed cycles by delay categories (1 week,

2 weeks, 3 weeks, 4 weeks and >4 weeks).

Number of patients with a dose delay due to COVID-19 pandemic will be summarized.

All melflufen and dexamethasone administration details will be presented in the respective listings.

7.9.2 ADVERSE EVENTS

All AE summaries will be presented based on the safety analysis set by cohort and overall.

All AEs will be coded using the MedDRA (version 24.0 or higher), for toxicity assessment the

National Cancer Institute Common Toxicity Criteria Adverse Event (NCI CTCAE) version 4.03

will be used.

The summaries of AEs will be based on treatment-emergent adverse events (TEAEs).

TEAEs are defined as AEs that start on or after the first day of study treatment (the earliest of

melflufen and dexamethasone start date) administration and within 30 days after the last

administration of study treatment (the latest of melflufen and dexamethasone end date), or before

start of subsequent anticancer treatment (whichever occurs first) or that worsen on or after the first

day of study treatment.

An overall summary of AEs will be presented. It will include the number and percentage of patients

(as well as total event count) with at least one pre-treatment condition (started prior to the first

dose of melflufen and/or dexamethasone), patients with at least one TEAE, patients with at least

one grade 3, grade 4 and grade 3/4 TEAE, patients with at least one serious TEAE, and patients

with TEAEs leading to death.

The overall summary will include the treatment related TEAEs analyzed separately for treatment

related TEAEs (melflufen and/or dexamethasone related), melflufen related TEAEs, and

dexamethasone related TEAE. It will include the number and percentage of patients (as well as

total event count) with each corresponding treatment related TEAEs; patients with grade 3, grade

CONFIDENTAL


4 and grade 3/4 TEAEs; This summary will include the number (%) of patients with study

treatment related serious TEAEs as well as melflufen-related serious TEAEs, and dexamethasone

related serious TEAE separately along with the number (%) of patients with respective treatment

related TEAEs leading to death. In addition the number and percentage of patients with TEAEs

leading to dose reduction, dose held and dose discontinuation will be presented for overall

(melflufen and/or dexamethasone), and separately for melflufen and dexamethasone.

The number and percentage of patients experiencing TEAEs, as well as total event count (except

for summaries by toxicity grade), will be summarized by MedDRA SOC and PT for:

• TEAEs

• Non-serious TEAEs

• Treatment-related (related to melflufen and/or dexamethasone) TEAEs

Melflufen-related TEAEs

• Dexamethasone-related TEAEs

Serious TEAEs

• Treatment-related serious TEAEs

Melflufen-related serious TEAEs

Dexamethasone-related serious TEAEs

• TEAEs by CTCAE toxicity grade

• Treatment related (related to melflufen and/or dexamethasone) TEAEs by CTCAE toxicity

grade

Melflufen-related TEAEs by CTCAE toxicity grade

• Dexamethasone-related TEAEs by CTCAE toxicity grade

• Serious TEAEs by CTCAE toxicity grade

Treatment-related serious TEAEs by CTCAE toxicity grade

• Melflufen-related serious TEAEs by CTCAE toxicity grade

• Dexamethasone-related serious TEAEs by CTCAE toxicity grade

• TEAEs resulting in any treatment modification (hold, reduction, delay, interruption and

discontinuation) for any study drug and also separately for melflufen and dexamethasone

The number and percentage of patients with grouped AEs – TEAEs defined as follows:

• Thrombocytopenia (SMQ "Haematopoietic thrombocytopenia" – Broad scope)


Neutropenia (PTs: "Neutropenia", "Febrile neutropenia", "Neutrophil count decreased",
 "Neutropenic sepsis", "Neutropenic infection", "Cyclic neutropenia", "Band neutrophil
 count decreased", "Band neutrophil percentage decreased", "Neutrophil percentage
 decreased", "Agranulocytosis", "Granulocyte count decreased", "Granulocytopenia")

- Anemia (standardized MedDRA query (SMQ) "Haematopoietic erythropenia" Broad scope)
- Myelodysplastic syndrome (PTs: "5q minus syndrome", "Chronic myelomonocytic leukemia", "Myelodysplastic syndrome", "Myelodysplastic syndrome transformation", "Myelodysplastic syndrome unclassifiable", "Refractory anemia with an excess of blasts", "Refractory anemia with ringed sideroblasts", "Refractory cytopenia with multilineage dysplasia", "Refractory cytopenia with unilineage dysplasia", "Sideroblastic anemia")
- Second primary malignancies ((SMQ "Malignant or unspecified tumours" and HLT "Myelodysplastic syndromes"), excluding HLGT "Plasma cell neoplasms")
- Febrile neutropenia (PT "Febrile neutropenia")
- Infections ( SOC "Infections and infestations")
- Infective pneumonia broad scope (SMQ "Infective pneumonia")
- Infective pneumonia narrow scope (SMQ "Infective pneumonia" Narrow terms)
- Hemorrhage (SMQ "Haemorrhages" Narrow terms)
- Thrombocytopenia concomitant to hemorrhage: Hemorrhage with an onset date within ± 7 days of the onset and/or resolution date of a grade 3 or 4 thrombocytopenia. Grade 3/4 thrombocytopenia resolution date is to be identified based on the laboratory data as a first day when thrombocytopenia assessment is grade 2 or lower (grade ≤ 2 for toxicity "Platelet count decreased").
- Neutropenia concomitant to infection: Infection with an onset date within ± 7 days of the onset and/or resolution date of a grade 3 or 4 neutropenia. Grade 3/4 neutropenia resolution date is to be identified based on the laboratory data as a first day when neutropenia assessment is grade 2 or lower (grade ≤ 2 for toxicity "Neutrophil count decreased").

The groups above will be summarized as a separate summaries for all by SOC, PT and all by SOC, PT, CTCAE toxicity grade analyses.

By SOC, PT grouped AE summaries will also be presented by cycle.


For by-cycle reporting, an AE is assigned to particular cycle if started at or after the date and time

of the study treatment (earliest of melflufen and dexamethasone administration at particular cycle)

administration at particular cycle and prior to the date of treatment administration in subsequent

cycle. If a patient discontinued somewhere in between the cycles, the AE is assigned to the cycle

in which the discontinuation has happened.

A patient reporting the same TEAE more than once will only be counted once when calculating

incidence:

• within a given SOC

within a given SOC and PT combination or MedDRA SMQ

The maximum CTCAE toxicity grade and strongest causal relationship to study treatment for the

event will be used in the incidence calculations.

TEAEs reported with a causality assessment of "Probably Related" and "Possibly Related" are to

be considered as "Related" for the analysis purposes. AEs having both onset and end dates missing

will be considered TEAEs; in case of a missing start date and a complete end date, the AE will be

considered a TEAE unless the end date is prior to the date of the first dose of study drug.

A separate summary will present the number and percentage of patients who died during the study

treatment period (between the first dose of treatment (the earliest of melflufen and dexamethasone

start date) and within 30 days after last dose of treatment (the latest of melflufen and

dexamethasone end date)) and on follow-up (more than 30 days after last treatment dose along

with the reason for deaths as well as the number of patients died within 60 days after first treatment

dose.

Any AEs related to COVID-19 will be presented as separate PTs specific to COVID-19 or

coronavirus.

Listings will be provided for patients experiencing AEs, SAEs, AEs resulting in drug withdrawal

and events with fatal outcome.

7.9.3 LABORATORY DATA

Laboratory data will be summarized for the safety analysis set by cohort and overall.

For the purposes of summarization in both the tables and listings, all laboratory values will be

converted to standardized units on Study Data Tabulation Model (SDTM) level. Hematology and

CONFIDENTAL


chemistry parameters will be summarized descriptively and changes from baseline to post-baseline

visits for each parameter will be presented. Urinalysis results will only be listed.

All the data from both scheduled and unscheduled time points will be included in the CTCAE

grade shift tables.

Shift tables for the change in CTCAE grade (with separate parts for decreased and increased grades) will be constructed for hematology and chemistry laboratory parameters, which have corresponding CTCAE grades to tabulate changes in NCI CTCAE (version 4.03) from baseline to

worst post-baseline on study (up to and including EOT visit) CTCAE grade. Number of patients

with grade 3 or higher toxicity will be summarized as counts and percentages by cycle. A separate

listing of all laboratory results corresponding to grade 3 or 4 will be provided.

The following list of parameters that will be presented in the toxicity grades laboratory tables:

Hematology

o Hemoglobin (increase, decrease)

Platelets (decrease)

White blood cells (WBC) (increase, decrease)

ANC (decrease)

Lymphocyte count (increase, decrease)

Serum Chemistry

Alanine aminotransferase (ALT) (increase)

Aspartate aminotransferase (AST) (increase)

Alkaline phosphatase (increase)

Total bilirubin (increase)

Creatinine (increase)

Calcium (increase, decrease)

Glucose (increase, decrease)

Albumin (decrease)

Potassium (increase, decrease)

Sodium (increase, decrease)

eGFR (decrease)

Review Status: FINAL

Version: 2.0 Version Date: 20JUL2021

For hemoglobin, ANC and platelet counts, CTCAE grade shift tables will also be additionally

presented by cycles. For this analysis by cycle, the maximum grade within each cycle is used for

analysis.

Time from the date of the first study drug dose (earliest of melflufen and dexamethasone

administration at particular cycle) in a particular cycle until the date of grade 3, grade 4 and grade

3/4 onset will be presented for each cycle for ANC and platelets. Time to onset of grade 3, grade

4 and grade 3/4 for ANC and platelets will also be presented overall (duration in days from the

treatment start until the date of grade 3, grade 4 and grade 3/4 respectively) and for completed

cycles.

For laboratory results reported with a prefix, for example "<" or ">", the value derived from the

reported results without a prefix will be analyzed.

A separate table will be produced for incidence of grade 4 neutropenia (grade 4 toxicity

"Neutrophil count decreased") and thrombocytopenia (grade 4 toxicity "Platelet count decreased")

based on laboratory data for completed cycles (cycles having a subsequent cycle available). The

table will include the number of patients dosed in each cycle, the number of patients dosed in

completed cycle, the number and percentage of patients with grade 4 neutropenia and grade 4

thrombocytopenia, number and percentage of patients with G-CSF (concomitant medication with

PT="Granulocyte Colony Stimulating Factor", "Filgrastim", "Pegfilgrastim", "Lenograstim",

"Lipegfilgrastim")) in each cycle, the number and percentage of patients with platelets transfusion

(concomitant medication with PT="Platelets") and erythrocytes transfusion (concomitant

medication with PT="Erythrocytes" and "Red blood cells") at each cycle.

Concomitant medication is assigned to the particular cycle if taken between the date of the

melflufen administration at a particular cycle and date of melflufen administration in subsequent

cycle. If patient discontinued somewhere in between the cycles concomitant medication is assigned

to the cycle in which the discontinuation has happened.

Another table will investigate the occurrence of grade 3 and 4 neutropenia and thrombocytopenia

leading to melflufen dose reduction per cycle, based on the laboratory data,

All laboratory data will be listed, including CTCAE toxicity grades and normal ranges. A listing

will be provided for urine pregnancy tests as well.

7.9.4 VITAL SIGNS

CONFIDENTAL 

Review Status: FINAL

Version: 2.0


Vital signs will be summarized using descriptive statistics for the safety analysis set by cohort and

overall.

Results and change from baseline to post-baseline time points for weight, blood pressure, pulse,

respiratory rate and temperature will be presented.

A patient data listing will be provided to document height, weight, and vital signs data.

7.9.5 PHYSICAL EXAMINATION

Physical examination will only be listed without a summary.

7.9.6 12-LEAD ELECTROCARDIOGRAM (ECG)

ECG data will be summarized for the safety analysis set by cohort and overall.

ECG data (heart rate, PR interval, QRS interval, QT interval, QTc-Fridericia (QTcF) interval, RR

interval) will be summarized using descriptive statistics, changes from baseline to EOT visit will

also be evaluated.

Shift tables from baseline (Normal/Abnormal-clinically significant/Abnormal – not clinically

significant) to EOT visit will be summarized for ECG interpretation data.

All ECG data collected will be presented in the listing.

7.9.7 CHEST X-RAY

Chest x-ray data will be listed without a summary.

7.10 OTHER ENDPOINTS AND ANALYSIS

7.10.1 ECOG

ECOG performance status will be summarized as counts and percentages using shift tables of

baseline versus worst performance status (largest ECOG value) during the study. Also, the number

of patients with decrease of  $\geq 1$  unit and  $\geq 2$  units respectively at the last available visit and at the

EOT visit will be summarized as counts and percentages to reflect the level of improvement in

ECOG values.

7.10.2 EGFR

The eGFR level at the start of each cycle and the changes from baseline over time will be

presented using descriptive statistics.

CONFIDENTAL


A patient data listing will be provided to document eGFR level by cycle.

8. INTERIM ANALYSIS

The interim analysis took place to support accelerated New Drug Application (NDA) submission

and was described in the separate interim SAP dated 28 June 2019.

An interim analysis for an interim clinical study report (iCSR) is planned when patients enrolled

in Cohort 1a and 1b have been followed until progression or up to at least 6 months after first dose.

The objective of this interim analysis is to evaluate PK, safety and efficacy in Cohort 1, moderately

impaired patients, to support regulatory submissions. As no inferential statistical analyses are

planned at the interim analysis, the interim has no impact on the statistical methods or presentation

of data for the final report.

9. DEVIATIONS FROM ANALYSIS AS DESCRIBED IN THE

**PROTOCOL** 

There are no deviations from analysis as described in the protocol.

10. PROGRAMMING SPECIFICATION

All outputs will be produced using SAS version 9.4 or a later version.

The margins should be at least 1.50 inches for the binding edge and 1.0 inches for all others.

In the top left portion of each table/listing, the protocol number will be presented. On the next line

a table/listing number followed by the title of the table/listing and population information will be

displayed. Horizontal lines will appear after the column heading of the table/listing. Footnotes will

be put under the main body of text at the bottom of the page. The source listing number will be

displayed for all tables. The SAS program name will appear bottom left in a string and the page

number will appear on the bottom right corner of each table/listing. The date and time of creation

of table/listing will appear bottom left under to the SAS program name line.

Courier New 8-point bold font will be used for all tables and listings. Usually, a landscape layout

is suggested for both tables and listings, but it is not mandatory. Any date information in the listing

will use the date9. format, for example, 07MAY2002.

Shells for unique tables and listings are provided in a separate Mock-Up TFLs document.

11. REFERENCES

CONFIDENTAL 


Rajkumar, S. V., J. L. Harousseau, B. Durie, et al. Consensus Recommendations for the Uniform Reporting of Clinical Trials: Report of the International Myeloma Workshop Consensus Panel 1. Blood. 2011; 117(18):4691-4695.

Brookmeyer R, Crowley J. A Confidence interval for the median survival time. Biometrics; 1982; 38: 29-41.

Palumbo A, et al. Revised International Staging System for Multiple Myeloma: A Report from International Myeloma Working Group. Journal of Oncology 2015. 33:26, 2863-2869.